CLINICAL TRIAL: NCT04674709
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Pharmacokinetics of Oleander 4X in Healthy Volunteers
Brief Title: Evaluation of the Safety and Pharmacokinetics of Oleander 4X in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avila Herbals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AH-O4X-11-2020-01
Record Dates: First submitted 2020-11-23; First posted 2020-12-19 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Flu-like Symptoms
Keywords: Flu-like symptoms; Avila Herbals; Phoenix Biotechnology

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled Phase I study that will investigate the safety and efficacy of OLEANDER 4X HPUS in Healthy Volunteers.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple: Triple (Participant, Care provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety of Oleander 4X HPUS (Placebo Comparator): : To evaluate the clinical safety of OLEANDER 4X HPUS in healthy volunteers relative to the control arm (placebo group).
  Interventions: Drug: Oleander 4X - single; Drug: Oleander 4X - double; Drug: Oleander 4X - quadruple; Drug: Placebo
- Pharmacokinetics evaluation of Oleander 4X HPUS (Experimental): To evaluate the pharmacokinetics of OLEANDER 4X HPUS versus placebo.
  Interventions: Drug: Oleander 4X - single; Drug: Oleander 4X - double; Drug: Oleander 4X - quadruple; Drug: Placebo

INTERVENTIONS:
Drug: Oleander 4X - single — Cohort 1 receive 4 doses of Oleander 4X in a 24-hour period for a period of seven days.
Drug: Oleander 4X - double — Cohort 2 receive 2 doses of either active drug or placebo 4 times per day in a 24-hour period for a period of seven days.
Drug: Oleander 4X - quadruple — Cohort 3 receive 4 doses of either active drug four times per day in a 24-hour period for a period of seven days.
Drug: Placebo — The placebo group receives 4 doses of placebo in a 24-hour period for a period of 7 days

SUMMARY:
The homeopathic medicine, Oleander 4X HPUS is indicated for temporary relief of symptoms associated with flu, such as muscle or body aches, headaches, chills and fever, cough, and congestion. The primary purpose of this study is to assess the safety of Oleander 4X HPUS in health male and female subjects compared to a placebo. This is a randomized, double blind, placebo-controlled Phase I Proof of Concept clinical trial to evaluate the safety and efficacy of OLEANDER 4X HPUS in Healthy Volunteers. Briefly, 45 Healthy volunteers who meet the eligibility criteria and agree to participation in the study will be placed on 1.0 mL of OLEANDER 4X HPUS, four-to-twelve times per day for seven days. For the pharmacokinetics study (cohorts 4-6), participants will take OLEANDER 4X HPUS at a prescribed dose one time.

The aim of the present study is to evaluate the safety of OLEANDER 4X HPUS. This real-world cohort provides a unique opportunity to study this medicine. This protocol outlines a study involving Healthy volunteers. Up to 45 volunteers will be recruited in specific health systems in the USA.

Second ARM, sub-study: As a second arm of this study, a random double blind, placebo-controlled pharmacokinetics study in healthy volunteers. Briefly, 15 healthy volunteers who meet the same eligibility criteria and agree to participation in the study will be placed on one, two, or 4 doses (1 mL per dose) of OLEANDER 4X HPUS one time.

This is effectively three ascending doses in 4 subjects on OLEANDER 4X HPUS, compared to the placebo (1 subject).

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the safety of OLEANDER 4X HPUS. This protocol outlines a study involving Healthy volunteers. Up to 45 volunteers will be recruited in the USA.

Second ARM, sub-study: As a second arm of this study, a random double blind, placebo-controlled pharmacokinetics study in healthy volunteers. Briefly, 15 healthy volunteers who meet the same eligibility criteria and agree to participation in the study will be placed on one, two, or 4 doses (1 mL per dose) of OLEANDER 4X HPUS one time.

This is effectively three ascending doses in 4 subjects on OLEANDER 4X HPUS, compared to the placebo (1 subject).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers.
* Subjects with no symptoms of respiratory illness such as fever, rhinorrhea, mild cough, sore throat, headache, fatigue, muscle pain, and malaise but with no shortness of breath.
* Male or non-pregnant female adult > 18 to 65 years of age at time of enrollment to include all races and ethnic minorities.
* Agree to the collection of blood specimens (for the pharmacokinetics study).
* Willingness of study participant to provide informed consent and accept randomization to any assigned treatment arm.
* Must agree not to enroll in another study of an investigational agent prior to Day 28 of study, unless hospitalized.

Exclusion Criteria:

* Signs of any respiratory distress or pulmonary infection defined as the need for non-invasive or invasive mechanical ventilator support, ECMO or shock requiring vasopressor support.
* Subjects with risk factors for severe disease (e.g. hypertension, diabetes, pulmonary, cardiovascular, renal, hepatic, neurologic disease or immune compromise, obesity, and pregnancy).
* Any previous history of clinically significant cardiovascular disease, including ventricular arrhythmias.
* Current use of cardiac glycosides or a known allergic reaction to cardiac glycosides or compounds of similar chemical or biologic composition.
* Any risk factors that can lead to severe COVID-19 including uncontrolled diabetes, hypertension, and systemic diseases including hepatic disease and renal insufficiency.
* Pregnancy or breastfeeding.
* Participation in any other clinical trial of an experimental treatment for COVID-19.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events, serious event, and any related reactions as assessed by CTCAE v5.0. | 1-7 days
proportion of subjects undergoing DLT events | 1-7 days
  Safety evaluation

SECONDARY OUTCOMES:
pharmacokinetic parameters - AreaUnderCUrve (AUCt) [Time Frame: 24 hours] | 0-24 hours
  AUCt plasma concentration of oleander (using Oleandrin as the marker) during 24 hours after administration.
half-life (t1/2) | 0-24 hours
  half-life (t1/2) of oleander extract (using Oleandrin as the marker) during 24 hours after administration.
maximum and minimum plasma concentration | 0-24 hours
  maximum and minimum plasma concentration of oleander extract (using Oleandrin as the marker) during 24 hours after administration.
total body clearance (Cltot) | 0-24 hours
  total body clearance (Cltot) of oleander extract (using Oleandrin as the marker) during 24 hours after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa G Obiso, PhD, Study Director — Avila Herbals
Locations (1):
- Dr. William Ball offices, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No